CLINICAL TRIAL: NCT04812379
Title: Abilify Prolonged Release Aqueous Suspension for Intramuscular Injection Specified Drug-use Results Survey (Prevention of Recurrence/relapse of Mood Episodes in Bipolar I Disorder)
Brief Title: Specified Drug-use Survey on Abilify Prolonged Release Aqueous Suspension for IM Injection (Prevention of Relapse of Mood Episodes in BP)
Status: Completed | Type: Observational
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 031-101-00461
Record Dates: First submitted 2021-03-16; First posted 2021-03-23 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Bipolar Disorder I
MeSH Terms: interventions — Injections, Intramuscular; Aripiprazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Abilify prolonged release aqueous suspension for IM injection (Aripiprazole) — The usual dose in adults is 400 mg of aripiprazole administered intramuscularly in the gluteal or deltoid muscle as a single dose once every 4 weeks. The dose may be decreased to 300 mg based on the patient's symptoms and tolerability.

SUMMARY:
To investigate the safety for an observation period of 52 weeks with use of Abilify prolonged release aqueous suspension for intramuscular (IM) injection in patients with bipolar I disorder for prevention of recurrence/relapse of mood episodes in the routine clinical setting. The early stage safety after the switching from oral aripiprazole to this IM injection is investigated including extrapyramidal syndrome and malignant syndrome. Information regarding efficacy is collected as well.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* patients with a known hypersensitivity to aripiprazole

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in Japan with bipolar I disorder who are planned to be newly started on Abilify prolonged release aqueous suspension for IM injection, switching from oral aripiprazole for the purpose of prevention of recurrence/relapse of mood episodes
Sampling Method: Non-Probability Sample
Enrollment: 535 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Safety Information (Adverse Event) | 52 weeks from the start date of Abilify prolonged release aqueous suspension for IM injection therapy
  Any untoward medicinal occurrence in a patient or clinical study subject administered a Medicinal Product and which does not necessarily have a causal relationship with this treatment (ICH-E2A Guideline).
  An Adverse Event can therefore be any unfavorable and unintended sign (e.g. abnormal laboratory finding), symptom, or disease temporally associated with the use of a Medicinal Product (Abilify Prolonged Release Aqueous Suspension), whether or not it is considered causally related to the Medicinal Product.
Number of Special Situations (e.g. Maternal (pregnancy and breastfeeding) exposure, paternal (via semen) exposure or Overdose/Incorrect dosage) | 52 weeks from the start date of Abilify prolonged release aqueous suspension for IM injection therapy
  Collecting any Situations related to the use of an Otsuka product which may or may not be associated with an adverse event:
  * Maternal (pregnancy and breastfeeding) or paternal (via semen) exposure;
  * Exposure during breastfeeding;
  * Overdose/Incorrect dosage, misuse, abuse (e.g. patient sharing products);
  * Medication errors (e.g. patient took wrong dose);
  * Lack of therapeutic efficacy (e.g. the product doesn't work);
  * Occupational exposure (e.g.: nurse administering the product is exposed);
  * Cases of suspected transmission of infectious agents;
  * Use of suspected or confirmed falsified product(s) or quality defect of the product(s);
  * Withdrawal reactions;
  * Accidental exposure (e.g.: child takes parent's product);
  * Drug-drug/drug-food interactions;
  * Unintentional use of product in a non-approved population (e.g.: pediatric or geriatric population);
  * Disease progression/exacerbation of existing disease
  (Safety Information)
Number of off-Label Use | 52 weeks from the start date of Abilify prolonged release aqueous suspension for IM injection therapy
  Collecting any type of off-Label Use that refers to situations where a product is intentionally used for a medical purpose not in accordance with the authorized product information. Off-label use also includes the intentional use in non-authorized population categories not indicated in the label.
  (Safety Information)
Incidence of Serious Adverse Event (e.g. resulting in death or life-threatening) | 52 weeks from the start date of Abilify prolonged release aqueous suspension for IM injection therapy
  Collecting the number of any adverse drug experience/event occurring at any dose which
  * results in death
  * is life-threatening
  * requires inpatient hospitalization or prolonged of existing hospitalization
  * results in persistent or significant disability or incapacity
  * is a congenital anomaly/birth defect
  * is medically significant.
  (Safety Information)
Incidence of Non-serious Adverse Events (i.e. all Adverse Events that do not meet the definition of a serious Adverse Event) | 52 weeks from the start date of Abilify prolonged release aqueous suspension for IM injection therapy
  Collecting the number of non-serious Adverse Events
  (Safety Information)

SECONDARY OUTCOMES:
Number of patients who recurrence/relapse of Mood Episodes | 52 weeks from the start date of Abilify prolonged release aqueous suspension for IM injection therapy
  Collecting the number of patients who recurrence/relapse of Mood Episodes (Efficacy Information)

CONTACTS AND LOCATIONS:
Overall Officials: Yasuhiko Fukuta, PhD, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Pharmacovigilance Department, Osaka, Osaka, Japan